CLINICAL TRIAL: NCT06996132
Title: A Phase 2 Clinical Study of CD20×CD3 Bispecific Antibody-Based Salvage Therapy Followed by CAR-T With or Without ASCT in R/R Aggressive B-Cell Lymphoma
Brief Title: Bispecific Antibody-Based Salvage Therapy Followed by CAR-T ± ASCT in R/R Aggressive B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025054
Record Dates: First submitted 2025-05-20; First posted 2025-05-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory Aggressive B-cell Lymphoma
Keywords: Glofitamab; CAR T-cell therapy; autologous stem cell transplantation
MeSH Terms: conditions — Recurrence | interventions — glofitamab; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glofitamab-based therapy followed by CAR-T ± ASCT (Experimental): Subjects will receive two cycles of glofitamab-based therapy, followed by either CAR-T cell therapy alone or in combination with ASCT.
  Interventions: Drug: Glofitamab; Drug: Chimeric Antigen Receptor T Cells (CAR-T)

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is administered as monotherapy or in combination with investigator-selected agents (including but not limited to chemotherapy, ADCs, BTK inhibitors, etc.) for 2 cycles.
Drug: Chimeric Antigen Receptor T Cells (CAR-T) — After two cycles of glofitamab-based salvage therapy, single-target or dual-target CAR-T cells directed against CD19, CD20, and/or CD22 are infused following lymphodepleting (fludarabine + cyclophosphamide) or myeloablative conditioning, at a dose of 2-4 × 10⁶/kg.

SUMMARY:
This study consists of two sequential treatment phases. In the first phase, patients with r/r aggressive B-NHL receive two cycles of glofitamab ± investigator-selected agents. In the second phase, patients eligible for CAR-T monotherapy undergo FC lymphodepletion followed by CAR-T infusion (2-4×10⁶/kg), while those eligible for CAR-T+ASCT receive conditioning chemotherapy with PBSC reinfusion on day 0 and CAR-T administration (2-4×10⁶/kg) on day +3 (±1). Patients demonstrating Deauville 4-5 or ctDNA positivity at day 28 post-CAR-T infusion subsequently receive four cycles of glofitamab consolidation therapy.

DETAILED DESCRIPTION:
The study comprises two sequential treatment phases. In the first phase, eligible patients with r/r aggressive B-NHL receive 2 cycles of glofitamab ± X regimen (where X includes but is not limited to chemotherapy, antibody-drug conjugates, or small-molecule targeted agents, selected at the investigator's discretion). Peripheral blood lymphocyte apheresis is performed prior to initial glofitamab administration unless clinically contraindicated, with hematopoietic stem cell mobilization and collection timed per investigator assessment to achieve minimum required yields of ≥3×10⁸/kg mononuclear cells and ≥2×10⁶/kg CD34+ cells.

Patients successfully completing phase 1 proceed to phase 2 treatment. In the CAR-T alone cohort, patients receive FC lymphodepleting therapy (days -5 to -3) followed by CAR-T cell infusion (2-4×10⁶/kg) on day 0. The CAR-T+ASCT cohort undergoes conditioning chemotherapy (regimen determined by investigator) with autologous PBSC reinfusion on day 0 and CAR-T cells (2-4×10⁶/kg) administered on day +3 (±1 day).

At day 28 post-CAR-T infusion, patients demonstrating PET-CT Deauville scores of 4-5 or ctDNA positivity initiate 4 cycles of glofitamab consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory aggressive B-cell lymphoma, including the following subtypes: diffuse large B-cell lymphoma (DLBCL), high-grade B-cell lymphoma (HGBL), or transformed large B-cell lymphoma.
2. Relapsed or refractory disease, meeting criteria for one of the following cohorts:

   Cohort 1 (Relapsed/Refractory Disease):
   1. ≥2 prior lines of therapy (including both anti-CD20 monoclonal antibody and anthracycline-based chemotherapy) with documented progression following last treatment; OR
   2. Failure of first-line immunochemotherapy (containing anti-CD20 antibody and anthracycline) defined by any of:

      * Relapse/progression within 12 months of treatment completion; OR
      * Progressive disease during first-line therapy; OR
      * Stable disease as best response after 4 cycles; OR
      * Partial response as best response after 6 cycles.

   Cohort 2 (Early Treatment Failure):
   * Persistent metabolic activity (Deauville 5) on PET-CT after 2 cycles of first-line immunochemotherapy; OR
   * Biopsy-proven residual disease following initial therapy.
3. Age ≥18 years and ≤65 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
5. Hematologic parameters at screening must meet the following (unless due to bone marrow involvement):

   * Absolute neutrophil count (ANC) ≥1×10⁹/L,
   * Platelet count (PLT) ≥75×10⁹/L.
6. Biochemical parameters at screening must meet the following:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN);
   * Total bilirubin (TBIL) ≤1.5×ULN (unless due to Gilbert's syndrome or non-hepatic causes);
   * Serum creatinine (Cr) ≤2×ULN OR creatinine clearance ≥40 mL/min.
7. Left ventricular ejection fraction (LVEF) within institutional normal range by echocardiography.
8. Baseline oxygen saturation >92% on room air.
9. Life expectancy ≥3 months as assessed by the investigator.

Exclusion Criteria:

1. Confirmed primary central nervous system lymphoma;
2. Prior autologous or allogeneic hematopoietic stem cell transplantation;
3. Active HBV or HCV infection, defined as HBV-DNA or HCV-RNA levels above the upper limit of detection.
4. Uncontrolled comorbidities include infectious diseases, cardiovascular/cerebrovascular disorders, coagulopathies, and connective tissue diseases.
5. History of epilepsy or other central nervous system disorders;
6. Pregnancy or lactation;
7. HIV infection;
8. History of other malignancies unless:

   1. Disease-free for ≥5 years, or
   2. Previously cured of the following:

      * Non-melanoma skin cancers (basal cell carcinoma, squamous cell carcinoma, or related localized cutaneous malignancies)
      * Carcinoma in situ of cervix
9. Other conditions deemed ineligible by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate after CAR-T±ASCT | From CAR-T±ASCT administration until 1 year post-treatment
  The complete response (CR) rate after CAR-T±ASCT is defined as the proportion of subjects achieving CR following CAR-T with or without ASCT.

SECONDARY OUTCOMES:
overall response rate after CAR-T±ASCT | From CAR-T±ASCT administration until 1 year post-treatment
  The overall response rate (ORR) after CAR-T±ASCT is defined as the proportion of subjects achieving CR or partial response (PR) following CAR-T with or without ASCT.
complete response rate before CAR-T±ASCT | From the initiation of glofitamab-based therapy until ≤14 days prior to the start of FC lymphodepleting therapy or myeloablative conditioning.
  The complete response rate before CAR-T±ASCT is defined as the proportion of subjects achieving CR on the last assessment before CAR-T ± ASCT.
overall response rate before CAR-T±ASCT | From the initiation of glofitamab-based therapy until ≤14 days prior to the start of FC lymphodepleting therapy or myeloablative conditioning.
  The overall response rate (ORR) before CAR-T±ASCT is defined as the proportion of subjects achieving CR or PR on the last assessment before CAR-T ± ASCT.
progression free survival-total (PFS-t） | through 2 years after initiation of study treatment
  PFS-t is measured from initiation of glofitamab-based therapy until disease progression, relapse, or death from any cause.
progression free survival-CART (PFS-c） | through 2 years after initiation of study treatment
  PFS-c is measured from initiation of CAR-T±ASCT therapy until disease progression, relapse, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China